CLINICAL TRIAL: NCT05357066
Title: Nitrous Oxide as Treatment for Fibromyalgia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB20-1169
Record Dates: First submitted 2021-11-09; First posted 2022-05-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Central Neuropathic Pain
Keywords: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Endothelium-Dependent Relaxing Factors; Inhalation; Nitrous Oxide; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a treatment group schedule, group-1 (nitrous, placebo), or group-2 (placebo, nitrous). Dosing consists of 50% Nitrous oxide in oxygen mixture (FiO2 0.5) vs placebo (oxygen-air mixture FiO2 ≈0.3).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and assessor blinded to study group assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment; Nitrous Oxide 50% (Active Comparator): A single 60-minute session of inhaled 50% nitrous oxide.
  Interventions: Drug: Nitrous oxide gas for inhalation
- Control; Oxygen-air mixture (Placebo Comparator): A single 60-minute session of inhaled Oxygen-air mixture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrous oxide gas for inhalation — Administration of inhaled 50% nitrous oxide in oxygen (FiO2 0.5) will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Other Names: Nitrous Oxide; Nitrous; N2O; Laughing gas
  Arms: Treatment; Nitrous Oxide 50%
Drug: Placebo — Administration of the placebo (oxygen-air mixture [FiO2 ≈0.3]), will be under the direct supervision of a licensed practitioner who is experienced in the use and administration of the study drug, and is familiar with the indications, effects, dosages, methods, and frequency and duration of administration, and with the hazards, contraindications, and side effects and the precautions to be taken (MD, or CRNA); with study patient monitoring of pulse oximetry, heart rate, respiratory, non-invasive blood pressure, and end-tidal carbon dioxide.
  Other Names: Sham
  Arms: Control; Oxygen-air mixture

SUMMARY:
The purpose of this study is to explore a potential role of nitrous oxide in treating pain associated with fibromyalgia.

DETAILED DESCRIPTION:
Investigators are conducting this trial to determine the efficacy of nitrous oxide on fibromyalgia, a chronic, debilitating, disorder typified by widespread musculoskeletal pain, accompanied by symptoms of fatigue, affected sleep, memory issues, and mood disorders.

Studies suggests that the chronic widespread pain seen in fibromyalgia patients has a neurogenic origin. Higher levels of ascending pathway neurochemicals, including nerve growth factor, substance P, and brain derived neurotrophic factor, are present in the cerebrospinal fluid (CSF) of fibromyalgia patients when compared to healthy controls. In addition, glutamate levels can be elevated in both the CSF and brain of fibromyalgia patients. Glutamate may play a central role, by acting on the NMDA-receptors to increase the central amplification of pain perception, which is thought to manifest as allodynia and hyperalgesia in fibromyalgia patients. NMDA-receptors are thus an attractive target for fibromyalgia therapeutic drug development.

In four other randomized controlled trial(s) to evaluate ketamine an NMDA-receptor antagonist; two demonstrated an acute reduction in VAS pain scores (20- to -25 points) 90- to 120-minutes following IV ketamine 0.3 mg/kg compared with placebo; while the other two using different drug concentrations and dose regimen (0.3 mg/kg over 30 minutes and 0.5 mg/kg for 3 hours) showed a 0.5- to 0.9-point reduction in pain scores (10-cm VAS) at 90 to 180 minutes following IV ketamine compared with placebo. Although all four trials demonstrated significant acute pain improvement during and immediately following the infusions, there were no sustained improvements.

Given nitrous oxide is another drug with known NMDA-receptor antagonism, this trial will evaluate the efficacy of inhaled 50% nitrous oxide compared to placebo (oxygen-air mixture). Study participants with a clinical diagnosis of fibromyalgia, meeting 2016-Fibromyalgia Diagnostic Criteria (2016-ACR) and neuropathic pain criterion will be randomly assigned to receive two, 60-minute inhalation sessions (50% nitrous oxide and placebo).

Treatment outcomes will be monitored using diagnostic tools measuring functionality, pain, and mood:

* Numeric Pain Rating Scale (NPRS)
* Revised Fibromyalgia Impact Questionnaire (FIQR)
* Patients Global Impression of Change Scale (PGIC)
* Hospital Anxiety and Depression Scale (HADS)
* Computerized Adaptive Test-Mental Health (CAT-MH)

ELIGIBILITY:
Inclusion Criteria:

* 2016 American College of Rheumatology Revised criteria for fibromyalgia (2016-ACR)
* Subjects 18 -75 years of age.
* Self-reported pain of at least 4 on the Numeric Pain Rating Scale (NPRS) at screening and baseline.
* Subject receives and agrees to remain on their stable fibromyalgia treatment plan established at least 4 weeks prior to dosing. Stable means no change in dose or any pain medication.
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments
* If currently on psychotherapy, it must have been maintained at the same frequency for 4 weeks prior to treatment.

Exclusion Criteria:

* Unstable doses of allowed antidepressants or muscle relaxants or dosages for any other medical condition.
* Pain due to concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, or other chronic widespread pain condition(s) that may confound fibromyalgia pain.
* Psychiatric or cognitive disorder (e.g., current schizophrenia, severe depression, suicidal ideation, dementia, etc.) that the investigator or sponsor considers significant for this study.
* Clinically significant alcohol or other substance abuse within the last 2 years, in the opinion of the investigator.
* Current or recent history of medically inappropriate or illegal use of drugs of abuse including benzodiazepines, opiates, cocaine, cannabinoids, and amphetamines.
* Current treatment with N-methyl-D-aspartate receptor (NMDAR) ligands including ketamine, amantadine, dextromethorphan, memantine, methadone, or dextropropoxyphene.
* Subjects who are pregnant, breast feeding, or planning to become pregnant during the course of the study and for 28 days after the final administration of investigational product.
* Any other serious medical condition affecting heart, lung or any other organ system.
* Any impairment, activity or situation that in the judgment of the investigator would prevent satisfactory completion of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Monitor changes in NPRS score | Over 8-weeks from baseline (length of study participation)
  Monitoring changes in 'Numeric Pain Rating Scale' (NPRS) diagnostic score to determine effectiveness a 60-minute session of inhaled 50% nitrous oxide vs placebo has on symptoms associated with fibromyalgia.
  The NPRS is a validated self-report diagnostic asking patients to indicate the intensity of current, best, and worst pain levels over the past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable).
  Response and remission will be based on a 30% improvement in average daily mean (max and min) NPRS score.

SECONDARY OUTCOMES:
Changes in FIQR | Over 8-weeks from baseline (length of study participation)
  Evaluation of response and remission will be based on 'Fibromyalgia Impact Questionnaire-Revised' (FIQR).
  This validated self-report diagnostic contains 21-questions to rate fibromyalgia effects over the prior 7-days.
  Domain 1: 9-questions rating function: 'No difficulty = 0' to 'Very difficult = 10' Domain 2: 2-questions rating overall impact: 'Never = 0' to 'Always = 10' Domain 3: 10-questions rating symptom intensity: 'None = 0' to 'Worst = 10'
  * First: Sum the scores for each of the 3 domains (function, overall, and symptoms).
  * Second: Divide domain 1 score by 3, leave domain 2 score unchanged, and divide domain 3 score by 2.
  * Third: Add the 3 resulting domain scores to obtain the total FIQR score.
Changes in Global Impression of Change Scale | Over 8-weeks from baseline (length of study participation)
  The Global Impression of Change Scale (PGI-C), a two question, self-report diagnostic evaluating the patients belief of treatment efficacy.
  - Patients rate their neuropathic pain ['No pain = 0' to 'Worst = 10'], and evaluate treatment effectiveness ['Very Much Improved'; 'Much Improved'; 'Minimally'; 'Improved'; 'No Change'; 'Minimally Worse'; 'Much Worse'; 'Very Much Worse']
Computerize Adaptive Testing - Mental Health (CAT-MH) measurements | Over 8-weeks from baseline
  This CAT-MH is a validated self-reporting diagnostic that adaptively selects a small optimal set of items from a large bank of approximately 1,500 items, targeted to individuals current or historical level of severity and likelihood of 'depression'.
  Generated scores include severity and liklihood percentile:
  depression = (%) normal, mild, moderate, severe
Hospital Anxiety and Depression Scale | Over 8-weeks from baseline (length of study participation)
  The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire comprising of 14-questions (7-anxiety and 7-depression), with response scores ranging: '0' to '3'
  * Sum Depression scores = 0 to 21
  * Sum Anxiety scores = 0 to 21
  Score range for each item (depression and anxiety):
  0-7 = Normal 8-10 = Borderline abnormal (mild) 11-14 = Abnormal (moderate) 15-21 = Severe

OTHER OUTCOMES:
Adverse events | Over 8-weeks (length of study participation)
  AEs such as nausea and vomiting; or any other AEs determined probably, possibly, or unrelated to the study intervention.
  Study patient safety is monitored by the investigators (MD) with experience in critical care anesthesia, as well as an experienced clinical research team responsible for recording and reporting events.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, MSc, Principal Investigator — University of Chicago, Department of Anesthesia and Critical Care
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold LM, Clauw DJ, Dunegan LJ, Turk DC; FibroCollaborative. A framework for fibromyalgia management for primary care providers. Mayo Clin Proc. 2012 May;87(5):488-96. doi: 10.1016/j.mayocp.2012.02.010. PMID 22560527
- [Background] Clauw DJ, Arnold LM, McCarberg BH; FibroCollaborative. The science of fibromyalgia. Mayo Clin Proc. 2011 Sep;86(9):907-11. doi: 10.4065/mcp.2011.0206. PMID 21878603
- [Background] Sorensen J, Bengtsson A, Backman E, Henriksson KG, Bengtsson M. Pain analysis in patients with fibromyalgia. Effects of intravenous morphine, lidocaine, and ketamine. Scand J Rheumatol. 1995;24(6):360-5. doi: 10.3109/03009749509095181. PMID 8610220
- [Background] Sorensen J, Bengtsson A, Ahlner J, Henriksson KG, Ekselius L, Bengtsson M. Fibromyalgia--are there different mechanisms in the processing of pain? A double blind crossover comparison of analgesic drugs. J Rheumatol. 1997 Aug;24(8):1615-21. PMID 9263160
- [Background] Noppers I, Niesters M, Swartjes M, Bauer M, Aarts L, Geleijnse N, Mooren R, Dahan A, Sarton E. Absence of long-term analgesic effect from a short-term S-ketamine infusion on fibromyalgia pain: a randomized, prospective, double blind, active placebo-controlled trial. Eur J Pain. 2011 Oct;15(9):942-9. doi: 10.1016/j.ejpain.2011.03.008. Epub 2011 Apr 11. PMID 21482474
- [Background] Graven-Nielsen T, Kendall SA, Henriksson KG, Bengtsson M, Sorensen J, Johnson A, Gerdle B, Arendt-Nielsen L. Ketamine reduces muscle pain, temporal summation, and referred pain in fibromyalgia patients. Pain. 2000 Apr;85(3):483-491. doi: 10.1016/S0304-3959(99)00308-5. PMID 10781923
- [Background] Jevtovic-Todorovic V, Todorovic SM, Mennerick S, Powell S, Dikranian K, Benshoff N, Zorumski CF, Olney JW. Nitrous oxide (laughing gas) is an NMDA antagonist, neuroprotectant and neurotoxin. Nat Med. 1998 Apr;4(4):460-3. doi: 10.1038/nm0498-460. PMID 9546794
- [Background] Nagele P, Metz LB, Crowder CM. Nitrous oxide (N(2)O) requires the N-methyl-D-aspartate receptor for its action in Caenorhabditis elegans. Proc Natl Acad Sci U S A. 2004 Jun 8;101(23):8791-6. doi: 10.1073/pnas.0402825101. Epub 2004 May 24. PMID 15159532